CLINICAL TRIAL: NCT00759434
Title: A Dual Centre, Randomised Controlled Trial of the Clinical and Cost Effectiveness of Endovenous Laser Therapy (EVLT) in the Treatment of Varicose Veins and Venous Ulcers
Brief Title: A New Method of Surgically Treating Varicose Veins and Venous Ulcers - a Study to Assess Clinical and Economic Value
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hull University Teaching Hospitals NHS Trust (Other Government)
Collaborators: University of Hull (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HELP1
Record Dates: First submitted 2008-09-23; First posted 2008-09-25 (Estimated); Last update posted 2022-08-19 (Actual); Status verified 2022-08

CONDITIONS: Varicose Veins; Venous Insufficiency; Venous Ulceration
Keywords: Varicose veins; Chronic venous insufficiency; Venous ulceration; Surgery; Endovenous Laser
MeSH Terms: conditions — Varicose Veins; Venous Insufficiency; Varicose Ulcer

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Surgery (Active Comparator)
  Interventions: Procedure: Surgery - Saphenofemoral ligation, saphenous strip and avulsions
- EVLT (Experimental)
  Interventions: Procedure: EVLT

INTERVENTIONS:
Procedure: Surgery - Saphenofemoral ligation, saphenous strip and avulsions — Patients undergo Saphenofemoral ligation, inversion stripping of the Long Saphenous Vein and avulsion of varicosities if necessary under a general anaesthetic.
  Arms: Surgery
Procedure: EVLT — Patients undergo endovenous laser treatment, using a 810nm laser aiming to occlude the incompetent long saphenous vein from the saphenofemoral junction to the knee. This may then be followed by ambulatory phlebectomy as appropriate. All procedures are to be performed under a local anaesthetic.
  Arms: EVLT

SUMMARY:
Varicose veins are a common problem, affecting up to a third of the western adult population. Most suffer with aching, discomfort, pruritis, and muscle cramps, whilst complications include oedema, eczema, lipodermatosclerosis, ulceration, phlebitis, and bleeding. This is known to have a significant negative effect on patient's quality of life (QoL).

Surgery has been used for many years, but it is known that there is a temporary decline in QoL post-op. This was demonstrated in our pilot study. Surgery leads to painful and prolonged recovery in some patients and has the risks of infection, haematoma and nerve injury.

Recurrence rates are known to be significant. Duplex of veins post surgery has demonstrated persistent reflux in 9-29% of cases at 1 year, 13-40% at 2 years, 40% at 5 years and 60% at 34 years.

26% of NHS patients were 'very dissatisfied' with their varicose vein surgery.

Newer, less invasive treatments are being developed. It would be advantageous to find a treatment that avoided the morbidity of surgery, one that could be performed as a day-case procedure under a local anaesthetic, a treatment that could offer lower recurrence rates and allow an early return to work. These should be the aims of any new treatment for varicose veins.

Endovenous Laser Treatment (EVLT) is performed under a local anaesthetic and uses laser energy delivered into the vein to obliterate it. The vein therefore need not be tied off surgically and stripped out.

The aim of this study is to compare the clinical, cost effectiveness and safety of Surgery and EVLT.

ELIGIBILITY:
Inclusion Criteria:

* Primary, symptomatic, varicose veins.
* Isolated Saphenofemoral junction (SFJ) incompetence leading to long saphenous (LSV) reflux on duplex ultrasound.
* LSV of 4mm diameter at the knee.
* Ability to give informed written consent.

Exclusion Criteria:

* Inability to give informed written consent.
* Symptomatic or complicated varicose veins not attributable to SFJ/LSV reflux.
* Evidence of deep venous reflux on duplex scan.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 280 (Actual)
Dates: Start 2004-03 (Actual); Primary Completion 2009-08 (Actual); Study Completion 2009-08 (Actual)

PRIMARY OUTCOMES:
Generic Quality of life - Short Form-36 | 1 week, 6 weeks, 3 months, 1 year, 2 years

SECONDARY OUTCOMES:
Disease Specific quality of life - Aberdeen Varicose Vein Questionnaire | 1 week, 6 weeks, 3 months, 1 year, 2 years
Generic quality of life - EuroQol | 1 week, 6 weeks, 3 months, 1 year, 2 years
Venous Clinical Severity Score | 3 months, 1 year, 2 years
Visual analogue pain scores | 1 week
Return to work and normal functioning | 1 week, 6 weeks
Would undergo EVLT again if necessary | 1 week, 6 weeks, 3 months, 1 year, 2 years
Complication rates | 1 week, 6 weeks, 3 months, 1 year, 2 years
Duplex and clinical assessment | 1 week, 6 weeks, 3 months, 1 year, 2 years
  A detailed clinical and duplex ultrasound assessment was undertaken to identify:
  The presence of residual or recurrent varicose veins (defined as clinically evident varicose veins of greater than 3mm in diameter present at 1 and 6 weeks (residual) or becoming evident only after 6 weeks (recurrent). This was irrespective of the presence or absence of symptoms.
  The pattern of underlying insufficiency on duplex giving rise to any clinically evident varicose veins or skin changes.
Cost Effectiveness | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Ian C Chetter, MBChB, Principal Investigator — University of Hull
Locations (1):
- Hull Royal Infirmary, Hull, East Yorkshire, United Kingdom

REFERENCES:
- [Background] Mekako AI, Hatfield J, Bryce J, Lee D, McCollum PT, Chetter I. A nonrandomised controlled trial of endovenous laser therapy and surgery in the treatment of varicose veins. Ann Vasc Surg. 2006 Jul;20(4):451-7. doi: 10.1007/s10016-006-9095-y. Epub 2006 Jun 27. PMID 16802211
- [Result] Carradice D, Mekako AI, Mazari FA, Samuel N, Hatfield J, Chetter IC. Clinical and technical outcomes from a randomized clinical trial of endovenous laser ablation compared with conventional surgery for great saphenous varicose veins. Br J Surg. 2011 Aug;98(8):1117-23. doi: 10.1002/bjs.7615. Epub 2011 Jun 3. PMID 21638277
- [Result] Carradice D, Mekako AI, Mazari FA, Samuel N, Hatfield J, Chetter IC. Randomized clinical trial of endovenous laser ablation compared with conventional surgery for great saphenous varicose veins. Br J Surg. 2011 Apr;98(4):501-10. doi: 10.1002/bjs.7394. Epub 2011 Jan 31. PMID 21283981
- [Derived] Mohamed AH, Howitt A, Rae S, Cai PL, Hitchman L, Wallace T, Nandhra S, Pymer S, Knighton A, Smith G, Chetter IC, Carradice D. Ten-year outcomes of a randomized clinical trial of endothermal ablation versus conventional surgery for great saphenous varicose veins. Br J Surg. 2024 Aug 2;111(8):znae195. doi: 10.1093/bjs/znae195. PMID 39162334
- [Derived] Wallace T, El-Sheikha J, Nandhra S, Leung C, Mohamed A, Harwood A, Smith G, Carradice D, Chetter I. Long-term outcomes of endovenous laser ablation and conventional surgery for great saphenous varicose veins. Br J Surg. 2018 Dec;105(13):1759-1767. doi: 10.1002/bjs.10961. Epub 2018 Aug 22. PMID 30132797
- [Derived] Carradice D, Wallace T, Gohil R, Chetter I. A comparison of the effectiveness of treating those with and without the complications of superficial venous insufficiency. Ann Surg. 2014 Aug;260(2):396-401. doi: 10.1097/SLA.0000000000000541. PMID 24424141
- [Derived] Carradice D, Mazari FA, Mekako A, Hatfield J, Allgar V, Chetter IC. Energy delivery during 810 nm endovenous laser ablation of varicose veins and post-procedural morbidity. Eur J Vasc Endovasc Surg. 2010 Sep;40(3):393-8. doi: 10.1016/j.ejvs.2010.04.010. Epub 2010 May 26. PMID 20510634